CLINICAL TRIAL: NCT04898530
Title: A Cross-sectional Assessment of Diet in Patients With IBD in Central Texas
Brief Title: Diet Patterns in IBD in Central Texas
Status: Suspended | Type: Observational
Why Stopped: interim analyses undeway
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Linda Anne Feagins, MD, Associate Professor, Director of Inflammatory Bowel Diseases Center, University of Texas at Austin
Other Study IDs: STUDY00000439
Record Dates: First submitted 2021-05-13; First posted 2021-05-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NO INTERVENTION — There is no intervention for this study.

SUMMARY:
The purpose of the study is to understand the diet patterns, preferences, and impact of diet on daily living in our patients with IBD in Central Texas.

ELIGIBILITY:
Inclusion Criteria:

* any patient 18years of age or older with inflammatory bowel disease

Exclusion Criteria:

* unwilling to participate
* diagnosis of IBD unable to be verified

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
diet patterns | 6 months
  diet descriptions, ASA24
diet preferences | 6 months
  via questionnaires
diet impact | 6 months
  various outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Medical School, UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided